CLINICAL TRIAL: NCT01202123
Title: Post Marketing Surveillance of MENOPUR
Status: Completed | Type: Observational
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: FE999906 CS10
Record Dates: First submitted 2010-09-03; First posted 2010-09-15 (Estimated); Last update posted 2014-02-21 (Estimated); Status verified 2014-02

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of highly purified (HP) menotrophine to Korean women.

ELIGIBILITY:
Inclusion Criteria:

* Anovulation in women (WHO group II)
* Controlled ovarian hyperstimulation cases for ART

Exclusion Criteria:

* Hypersensitivity to MENOPUR
* Pregnancy, lactation or contraindication to pregnancy
* Ovarian cysts not related to polycystic ovarian syndrome
* Abnormal uterine bleeding
* Tumors in uterus, ovaries and breasts
* Ovarian hyperstimulation syndrome
* Thromboembolism or history of it
* Infertile due to other reason than anovulation
* High FSH level indication primary ovarian failure

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Infertile women
Sampling Method: Probability Sample
Enrollment: 2501 (Actual)
Dates: Start 2008-12; Primary Completion 2013-11 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Number of follicles per cycle | Up to 6 weeks
  An ART cycle: From ovulation (number and size) to when chemical pregnancy test results are recorded

SECONDARY OUTCOMES:
Number of adverse events | Up to 6 weeks
  An ART cycle: From ovulation (number and size) to when chemical pregnancy test results are recorded

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (19):
- South Korea (19):
  - Busan Maria hospital, Busan, Busan
  - Daegu Maria, Daegu, Daegu
  - Daejeon Maria, Daejeon, Daejeon
  - Daejeon Seoul Women Hospital, Daejeon, Daejeon
  - Ellemedi Women Clinic, Daejeon, Daejeon
  - Miz Women's Hospital, Daejeon, Daejeon Metropolitan City
  - Seoul´s Women´s Hospital, Bucheon-si, Gyeonggi Province
  - Ilsan Maria Hospital, Ilsan, Gyeonggi Province
  - Incheon Seoul women Hospital, Incheon, Incheon
  - Premedi Women's Clinic, Kwangju, Kwangju Metropolitan City
  - Gumi CHA University Medical Center, Gumi, Kyoungbuk Province
  - Mama Papa & Baby Hospital, Ulsan, Kyoungnam Province
  - Cheil General Hospital & Women's Healthcare Center, Seoul, Seoul
  - Gangseo Mizmedi Hospital, Seoul, Seoul
  - Hamchoon women clinic, Seoul, Seoul
  - Maria Plus Hospital, Seoul, Seoul
  - Samsung Medical Center, Seoul, Seoul
  - Songnae Maria Hospital, Seoul, Seoul
  - Maria Hospital, Seoul, ´Shinseoul-dong, Dongdaemun-gu